CLINICAL TRIAL: NCT02076789
Title: Detect Long-term Complications After ICD Replacement: a Multicenter Italian Registry - DECODE Registry
Brief Title: DEtect Long-term Complications After icD rEplacement: a Multicenter Italian Registry
Acronym: DECODE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mauro Biffi (Other)
Responsible Party: Sponsor-Investigator, Mauro Biffi, Dirigente Medico di Cardiologia, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Other Study IDs: 72/2013/O/Oss
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Device Replacement; Device Upgrade; Long-term Postoperative Complications; Resource Consumption and Associated Costs After Device Replacement/Upgrade
Keywords: Device Replacement; Device Upgrade; Long-term Postoperative Complications; Resource consumption and associated costs after device replacement/upgrade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD generator replacement: Patients with standard indications to ICD generator replacement

SUMMARY:
This study has been designed to prospectively estimate long term complication rates (12-months and 5-years) in patients undergoing Implantable Cardioverter Defibrillator (ICD) replacement, with and without a planned transvenous lead addition for replacement or upgrade to a device capable of additional therapies; the study also evaluates the predictors of complications, the patient's management before and during the replacement procedure in clinical practice and the estimated costs related to the use of health care resources.

DETAILED DESCRIPTION:
Based on positive outcomes from numerous randomized, controlled trials, the implantable defibrillators have been included in the current European Society of Cardiology (ESC) and American College of Cardiology / American Heart Associations (ACC/AHA) guidelines as a standard of care in selected patients, and thus ICD use is currently increasing worldwide.

In the years after initial implantation, device replacement may become necessary for battery depletion or for upgrades to more complex multi-lead ICDs. The increase in generator or lead advisories and recalls contributes further to those patients considered for replacement.

The determination of procedural adverse events is complex, and requires monitoring of both short-term complications and long-term patient outcome.

Previous retrospective series have examined complications with ICD replacements. Moreover, the more recent REPLACE registry prospectively collected 6-month complication rates in patients undergoing pacemaker or ICD generator replacement at 72 private practice and academic sites in United States. This study examined a broad range of major and minor complications and found that ICD replacements were associated with a notable complication risk, particularly when a transvenous lead addition or revision was required.

Previous retrospective series have examined complications with ICD implantation in the Italian clinical practice, showing frequent interventions for system revision and demonstrating an association between adverse events and the complexity of the implanted device (i.e. Cardiac Resynchronization Therapy CRT-D versus single- or dual-chamber ICD). Moreover, it was shown that device replacement procedures are associated with significantly higher risk of infections.

Nonetheless, detailed data on the complications of ICD replacement in the current Italian clinical practice are unavailable.

This information would be particularly important because ICD replacement-related events may be associated not only with a worse clinical outcome, but also with incremental costs to the healthcare system.

The analysis of adverse events would permit to study new preventative strategies with significant clinical as well as financial benefits. Moreover, the quantification of the complication rate after ICD replacement would permit to estimate the actual long-term cost of ICD therapy, and to assess the impact of ICD longevity on the cost-effectiveness of the therapy.

This study has been designed to prospectively estimate long term complication rates (at 12-months and 5-years) in patients undergoing ICD generator replacement. The study also evaluates predictors of complications, patient's management before and during the replacement procedure in clinical practice and the estimated costs related to the use of health care resources.

All consecutive patients with standard indications to ICD generator replacement will be enrolled In this study. The decision to perform the generator replacement or to upgrade an existing device will be made according to the investigators' clinical assessment of their patient. The study do not mandate specific surgical or implantation techniques such as venous access, use of temporary pacemakers, or surgical site choices. Any commercially available generator or lead can be included.

Patients will be followed for a 60-month period with periodical in-hospital visits or remote ICD interrogations via remote patient monitoring (RPM) systems, according to the standard hospital practice and the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a CardiacResynchronizationTherapy-Defibrillator or single chamber/dual chambers ICD device (any commercially available generator or lead can be included).
* Patient with standard indications to ICD generator replacement according to the investigators' clinical assessment.
* Patient must be able to attend all required follow-up visits at the study center.

Exclusion Criteria:

* Patient is less than 18 years of age.
* Patient is unwilling or unable to sign an authorization to use and disclose health information or an Informed Consent.
* Patient life expectancy is less than 12 months.
* Patient is participating in another clinical study that may have an impact on the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing ICD generator replacement, with and without a planned transvenous lead addition for replacement or upgrade to a device capable of additional therapies (consecutive patients)
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Rate of complications associated with the ICD replacement / upgrade that occur during a period of 12 months | 12 months
  The primary outcome measure of this study is to estimate, at 12-months follow up, the percentage of subjects undergoing ICD generator replacement, with and without a planned transvenous lead addition for replacement or upgrade to a device capable of additional therapies, experiencing one of the pre-defined complications.

SECONDARY OUTCOMES:
Baseline patient's characteristics (clinical history and drug therapy) for subjects undergoing ICD replacement/upgrade | 60 months
  This secondary outcome measure of this study is to evaluate baseline patient's characteristics or variables of procedure's management as potential predictors of complications, that will be evaluated at 30 days, at 12 months and 60 months follow up
- Rate of complications associated with the ICD replacement / upgrade that occur during a very long-term period | 60 months
  This extends to 60 months the results obtained with the primary objective at 12 months
Long-term costs of ICD/upgrade procedure | 60 months
  This secondary outcome measure of this study is to evaluate resource consumption and associated costs in terms of devices, replacement/upgrade procedures , follow-up, post-replacement/upgrade management of complications and health care resources utilization.

CONTACTS AND LOCATIONS:
Locations (32):
- Italy (32):
  - Ospedale di Venere, Carbonara di Bari, Bari
  - A.O. "Papa Giovanni XXIII", Bergamo, BG
  - Ospedale di Bentivoglio, Bentivoglio, Bologna
  - Ospedale SS. Annunziata, Cento, Ferrara
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Ospedale "Maurizio Bufalini", Cesena, Forlì
  - Ospedale Maggiore, Lodi, LO
  - Ospedale Civile S.Agostino-Estense, Baggiovara, Modena
  - A.O.U.P. "Paolo Giaccone", Palermo, PA
  - Policlinico Universitario "Agostino Gemelli", Rome, RM
  - Ospedale Santa Maria alle Scotte, Siena, SI
  - Casa di Cura "Villa Verde", Taranto, TA
  - Ospedale "San Donato", Arezzo
  - Ospedale Maggiore, Bologna
  - Azienda Ospedaliera Universitaria , Policlinico Sant'Orsola, Bologna
  - Università Cattolica del Sacro Cuore, Campobasso
  - Ospedale Cuneo, Cuneo
  - Ospedale "San Giuseppe", Empoli
  - A.O.S.Anna, Ferrara
  - Ospedale "Morgagni-Pierantoni", Forlì
  - Ospedale "Padre Antero Micone" - Sestri Ponente, Genova
  - Ospedale della Misericordia, Grosseto
  - Clinica Mediterranea, Napoli
  - Ospedale Monaldi SUN, Napoli
  - A.O. Santa Maria della Misericordia, Perugia
  - Azienda Ospedali Riuniti Marche Nord, Pesaro
  - Ospedale "Santa Maria delle Croci", Ravenna
  - Ospedale Santa Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi, Rimini
  - Policlinico Casilino, Roma
  - A.O. San Giovanni di Dio e Ruggi di Aragona, Salerno
  - Ospedale Santa Maria di Cà Foncello, Treviso

REFERENCES:
- [Derived] Zoni-Berisso M, Martignani C, Ammendola E, Narducci ML, Caruso D, Miracapillo G, Notarstefano P, Carinci V, Pierantozzi A, Ciaramitaro G, Calo L, Zennaro M, Infusino T, Ferretti C, Sassone B, Licciardello G, Setti S, Terzaghi C, Malacrida M, Biffi M. Mortality after cardioverter-defibrillator replacement: Results of the DECODE survival score index. Heart Rhythm. 2021 Mar;18(3):411-418. doi: 10.1016/j.hrthm.2020.11.024. Epub 2020 Nov 27. PMID 33249200
- [Derived] Biffi M, Ammendola E, Menardi E, Parisi Q, Narducci ML, De Filippo P, Manzo M, Stabile G, Potenza DR, Zanon F, Quartieri F, Rillo M, Saporito D, Zaca V, Berisso MZ, Bertini M, Tumietto F, Malacrida M, Diemberger I. Real-life outcome of implantable cardioverter-defibrillator and cardiac resynchronization defibrillator replacement/upgrade in a contemporary population: observations from the multicentre DECODE registry. Europace. 2019 Oct 1;21(10):1527-1536. doi: 10.1093/europace/euz166. PMID 31209482
- [Derived] Zanon F, Martignani C, Ammendola E, Menardi E, Narducci ML, DE Filippo P, Santamaria M, Campana A, Stabile G, Potenza DR, Pastore G, Iori M, LA Rosa C, Biffi M. Device Longevity in a Contemporary Cohort of ICD/CRT-D Patients Undergoing Device Replacement. J Cardiovasc Electrophysiol. 2016 Jul;27(7):840-5. doi: 10.1111/jce.12990. Epub 2016 Jun 17. PMID 27094359
- [Derived] Diemberger I, Parisi Q, De Filippo P, Narducci ML, Zanon F, Potenza DR, Ciaramitaro G, Malacrida M, Boriani G, Biffi M. Detect Long-term Complications After ICD Replacement (DECODE): Rationale and Study Design of a Multicenter Italian Registry. Clin Cardiol. 2015 Oct;38(10):577-84. doi: 10.1002/clc.22440. Epub 2015 Aug 18. PMID 26282191